CLINICAL TRIAL: NCT06604000
Title: Goal Management Training (GMT) for Improvement of Cognitive Control Function After Acquired Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 62983
Record Dates: First submitted 2024-08-13; First posted 2024-09-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Acquired Brain Injury; Executive Function Disorder
Keywords: acquired brain injury; goal management training; executive function; cognitive control; GMT; cognitive rehabilitation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GMT Usual (+ GMT No Boost) (Active Comparator): Participants will receive Goal Management Training in groups of 4-6 patients, as implemented in a rehabilitation hospital setting (St. Olavs Hospital, Trondheim University Hospital). The standard treatment ("GMT Usual") consists of 10 sessions, delivered as 2 sessions a day, one day per week, over 5 weeks.
  Interventions: Behavioral: GMT Usual
- GMT Usual + GMT Boost (Experimental): Participants will receive Goal Management Training in groups of 4-6 patients, as implemented in a rehabilitation hospital setting (St. Olavs Hospital, Trondheim University Hospital). The standard treatment ("GMT Usual") consists of 10 sessions, delivered as 2 sessions a day, one day per week, over 5 weeks. After completion of the 10 GMT sessions and the first post-treatment assessment immediately after the main treatment period, the participants will receive an additional booster module ("GMT Boost") 3 months after the last ordinary GMT module - intended to facilitate a prolonged treatment response.
  Interventions: Behavioral: GMT Usual; Behavioral: GMT Boost
- GMT Usual + GMT Cuing (+ GMT No Boost) (Experimental): Participants will receive Goal Management Training in groups of 4-6 patients, as implemented in a rehabilitation hospital setting (St. Olavs Hospital, Trondheim University Hospital). The standard treatment ("GMT Usual") consists of 10 sessions, delivered as 2 sessions a day, one day per week, over 5 weeks. In this arm participants will also receive extended cuing through a smartphone application ("GMT Cuing") - intended to facilitate the effect of between-session tasks (homework) completed by the participants. These participants will, in addition to the standard treatment (as in "GMT Usual"), on a daily basis receive a message that says "STOP" as a reminder to do their home assignments. An sms with the the text "STOP" as a reminder everyday from the third session until the fifth session. The message is pseudorandomly sent on different timepoints ranging from 11am to 8pm, including in weekends.
  Interventions: Behavioral: GMT Usual; Behavioral: GMT Cuing
- GMT Usual + GMT Cuing + GMT Boost (Experimental): Participants will receive GMT Usual + GMT Cuing (see description above). In this arm, after completion of the 10 GMT sessions and the first post-treatment assessment immediately after the main treatment period, the participants will also receive an additional booster module ("GMT Boost") 3 months after the last ordinary GMT module - intended to facilitate a prolonged treatment response.
  Interventions: Behavioral: GMT Usual; Behavioral: GMT Cuing; Behavioral: GMT Boost

INTERVENTIONS:
Behavioral: GMT Usual — Participants will receive Goal Management Training in groups of 4-6 patients, as implemented in a rehabilitation hospital setting (St. Olavs Hospital, Trondheim University Hospital). The standard treatment ("GMT Usual") consists of 10 sessions, delivered as 2 sessions a day, one day per week, over 5 weeks.
Behavioral: GMT Cuing — The participants will receive extended cuing through a smartphone application ("GMT Cuing") - intended to facilitate the effect of between-session tasks (homework) completed by the participants. These participants will, in addition to the standard treatment (as in "GMT Usual"), on a daily basis receive a message that says "STOP" as a reminder to do their home assignments. An sms with the the text "STOP"; as a reminder everyday from the third session until the fifth session. The message is pseudorandomly sent on different timepoints ranging from 11am to 8pm, including in weekends.
  Arms: GMT Usual + GMT Cuing (+ GMT No Boost); GMT Usual + GMT Cuing + GMT Boost
Behavioral: GMT Boost — After completion of the 10 GMT sessions and the first post-treatment assessment immediately after the main treatment period, the participants will receive an additional booster module ("GMT Boost") 3 months after the last ordinary GMT module - intended to facilitate a prolonged treatment response.
  Arms: GMT Usual + GMT Boost; GMT Usual + GMT Cuing + GMT Boost

SUMMARY:
The goal of this clinical trial is to investigate predictors of treatment outcome, and the effect of individual treatment components of Goal Management Training (GMT) for improvement of cognitive control function in people with acquired brain injury (ABI).

Primary aim: To identify demographic, clinical and cognitive predictors of treatment response in Goal Management Training after acquired brain injury (ABI)?

Secondary aims: To investigate the effects of a) extended cuing (via a smartphone) and b) a booster module?

* All included participants will receive Goal Management Training in groups of 4-6 patients, as implemented in a rehabilitation hospital setting (St. Olavs Hospital, Trondheim University Hospital). The standard treatment ("GMT Usual") consists of 10 sessions, delivered as 2 sessions a day, one day per week, over 5 weeks.
* All participants will be asked to complete self-report measures and performance-based cognitive testing at baseline (T1), immediately after the main treatment period (T2), at 6 months (T3), and 1 year (T4) after treatment.
* After baseline assessment, 50% of participants will be randomized to receive extended cuing through a smartphone application ("GMT Cuing") - intended to facilitate the effect of between-session tasks (homework) completed by the participants. These participants will, in addition to the standard treatment, on a daily basis receive a message that says "STOP" as a reminder to do their home assignments.
* After completion of the 10 GMT sessions and the first post-treatment assessment immediately after the main treatment period, 50% of the participants will be randomized to receive an additional booster module ("GMT Boost") 3 months after the last ordinary GMT module - intended to facilitate a prolonged treatment response. The remaining 50% will receive no booster module ("GMT No Boost")
* Randomization will be carried out on treatment group-level (all patients in the same group receive the same treatment). The total anticipated sample size is N = 116 patients.
* The Global Executive Composite (GEC) score derived from BRIEF-A will be used as the primary outcome measure. A selection of other included measures will be used as secondary outcome measures.

DETAILED DESCRIPTION:
The Global Executive Composite (GEC) score derived from BRIEF-A will be used as the primary outcome measure. A selection of other included measures will be used as secondary outcome measures. Data will be analyzed based on an intention-to-treat approach. Penalized linear regression by the elastic net approach (a combination of the Lasso and Ridge regression approaches) will be used to identify demographic, clinical and cognitive predictors of outcome at 6 months after treatment (T3), which is the primary aim of the study. For the secondary aim of investigating the differences in outcome for primary and secondary outcomes between "GMT Cuing" and "GMT Usual", and between "GMT Boost" and "GMT No Boost", linear mixed models (LMMs) will be used. Data for all time points will be included, but of primary interest are differences at T2 (immediately after treatment) for assessing the effect of cuing, and at T3 (6 months after treatment) for the effect of boosting. The LMMs can account for within-subject correlations due to repeated measurements. In addition, the investigators will perform exploratory moderation and mediation analyses across both treatment groups. For the penalized regression models, complete case analyses will be performed as long as the number of missing observations is small. Otherwise, imputation will be considered, but imputation is not straightforward for variable selection models. Linear mixed models can handle missing data for the outcome variable. Considering multiple testing linked to several secondary outcomes, p-values will be interpreted with care rather than using a formal p-value adjustment. Results will be interpreted according to the magnitude of the group difference (effect size) as well as the p-values. Data will be analyzed using IBM SPSS, STATA and R.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 with acquired brain injury with no concomitant diseases minimum 12 months' post-injury/surgery, reporting cognitive control problems by structured interview or clinical performance measures.

Exclusion Criteria:

* Non-fluency in Norwegian Language
* Major psychiatric disorder or reported ongoing alcohol or substance abuse.
* Premorbid neurological disease or insult and/or comorbid neurological disease.
* Aphasia or other specified language problems causing potential communication problems.
* Impaired basic linguistic, mnemonic, motor, or perceptual function that can interfere with the ability to engage with training or estimated IQ < 85

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2029-12-18 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
The Global Executive Composite score from BRIEF-A | Baseline, Immediately after treatment, 6 months and 1 year after treatment
  Assessed with the Behavior Rating Inventory of Executive Function for Adults (BREIF-A), a 75 item questionnaire that that captures views of an adult's executive functions or self- regulation in his or her everyday environment. Items are rated on a 3-point scale (Never a problem - sometimes a problem - often a problem).
  Range:70-210. Higher score indicate greater executive dysfunction.

SECONDARY OUTCOMES:
Conners Continuous Performance Test -III (CPT-III) | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Wechslers Adult Inteligence Scale IV (WAIS-IV): Block Design | Baseline
Wechslers Adult Inteligence Scale IV (WAIS-IV): Matrix | Baseline
Wechslers Adult Inteligence Scale IV (WAIS-IV): Vocabulary | Baseline
Wechslers Adult Inteligence Scale IV (WAIS-IV): Similarities | Baseline
California Verbal Learning Test 2 (CVLT-2) | Baseline
Rey Complex Figure Test (Rey-O) | Baseline
Behavior rating Inventory of Executive function (BRIEF-A): significant other | Baseline, Immediately after treatment, 6 months and 1 year after treatment
D-KEFS: Tower | Baseline, Immediately after treatment, 6 months and 1 year after treatment
D-KEFS: Trail Making Test (TMT) | Baseline, Immediately after treatment, 6 months and 1 year after treatment
D-KEFS: Word Fluency | Baseline, Immediately after treatment, 6 months and 1 year after treatment
D-KEFS: Stroop Color-Word Interference Test | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Hopkins Symptom Checklist | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Achenbach System of Empirically Based Assessment (ASEBA): adult self-report | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Achenbach System of Empirically Based Assessment (ASEBA): adult behavior checklist (ABCL) | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Resilience Scale for Adults | Baseline, Immediately after treatment, 6 months and 1 year after treatment
The Metacognition questionnaire (MCQ-30) | Baseline, Immediately after treatment, 6 months and 1 year after treatment
SF-12 | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Pittsburg Sleep Quality Index | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Insomnia Severity Index | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Epworth Sleepiness Scale | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Fatigue Severity Scale | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Community Integration Questionnaire | Baseline, Immediately after treatment, 6 months and 1 year after treatment
Group Session Rating Scale (GSRS) | After each "GMT usual" treatment session (5 times throughout 5-weeks) and after the booster session ("GMT boost" at 3 months after last "GMT usual" session)
Week to week change rating scale ORS | After each "GMT usual" treatment session (5 times throughout 5-weeks) and after the booster session ("GMT boost" at 3 months after last "GMT usual" session)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Olsen, Principal Investigator — National Taiwan Normal University
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No
Individual patient data cannot be shared in this study due to laws and regulations in Norway.